CLINICAL TRIAL: NCT02905331
Title: A Phase 3, Multicenter, Randomized, Double-blind Placebo-controlled Study Evaluating the Efficacy and Safety of CNTO 1959 (Guselkumab) Delivered Via a SelfDose (TM) Device in the Treatment of Subjects With Moderate to Severe Plaque-Type Psoriasis
Brief Title: Efficacy and Safety Study of Guselkumab in the Treatment of Participants With Moderate to Severe Plaque-Type Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108203; CNTO1959PSO3006 (Other: Janssen Research & Development, LLC); 2016-002022-37 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Guselkumab: Placebo) (Experimental): Participants will receive 100 milligram (mg) guselkumab administered as a 100 milligram per milliliter (mg/mL) solution in a single-use prefilled syringe (PFS) assembled in a SelfDose device at Weeks 0, 4, 12, 20, and 28; liquid placebo for guselkumab 100 mg at Week 16 to maintain the study blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2 (Placebo: Guselkumab) (Experimental): Partcipants will receive placebo at Weeks 0, 4, and 12 followed by guselkumab 100 mg at Weeks 16, 20, and 28.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 100 mg of Guselkumab as 100 mg/mL solution via SelfDose device.
  Other Names: CNTO 1959
Drug: Placebo — Participants will receive matching placebo supplied in a PFS assembled in a SelfDose device.

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, pharmacokinetics, immunogenicity, usability, and acceptability of guselkumab delivered using SelfDose device in participants with moderate to severe plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* A woman of childbearing potential must have a negative urine pregnancy test (beta-human chorionic gonadotropin) at screening and at Week 0
* Before randomization, a woman must be either: a) Not of childbearing potential: premenarchal; postmenopausal (greater than [>] 45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle-stimulating hormone level (FSH) >40 International Units Per Liter [IU/L]); permanently sterile (example, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy, b) Of childbearing potential and practicing a highly effective method of birth control, consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: example, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal foam/gel/ film/cream/suppository (if available in their locale); male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence (when this is in line with the preferred and usual lifestyle of the participant)
* Agree not to receive a Bacillus Calmette Guerin (BCG) vaccination during the study, or within 12 months after the last administration of study drug
* Have a Psoriasis Area and Severity Index (PASI) greater than or equal to [>=] 12 at screening and at baseline
* Have an involved body surface area (BSA) >= 10 percent (%) at screening and at baseline

Exclusion Criteria:

* Has unstable cardiovascular disease, defined as a recent clinical deterioration (eg, unstable angina, rapid atrial fibrillation) in the last 3 months or a cardiac hospitalization within the last 3 months
* Has a history of lymphoproliferative disease, including lymphoma; a history of monoclonal gammopathy of undetermined significance (MGUS); or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy or splenomegaly
* Has a transplanted organ (with exception of a corneal transplant >3 months before the first administration of study drug)
* Has a nonplaque form of psoriasis (example, erythrodermic, guttate, or pustular)
* Has received any anti-tumor necrosis factor alpha (TNF-alpha) biologic therapy within 3 months before the first administration of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- United States (8):
  - Renstar Medical Research, Ocala, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - University of Pittsburgh Department of Dermatology, Pittsburgh, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island
  - Virginia Clinical Research, Norfolk, Virginia
- Canada (3):
  - Dr. Chih ho Hong Medical, Surrey, British Columbia
  - Dermatrials Research, Hamilton, Ontario
  - DermEdge Research, Mississauga, Ontario
- Poland (3):
  - Niepubliczny Zaklad Opieki Zdrowotnej Osteo-Medic s.c. Artur Racewicz i Jerzy Supronik, Bialystok
  - Szpital Uniwersytecki nr 1 im Dr A Jurasza, Bydgoszcz
  - Wromedica Irena Bielicka, Janusz Szczepanik S.C., Wroclaw

REFERENCES:
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Ferris LK, Ott E, Jiang J, Hong HC, Li S, Han C, Baran W. Efficacy and safety of guselkumab, administered with a novel patient-controlled injector (One-Press), for moderate-to-severe psoriasis: results from the phase 3 ORION study. J Dermatolog Treat. 2020 Mar;31(2):152-159. doi: 10.1080/09546634.2019.1587145. Epub 2019 Mar 19. PMID 30887876

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to guselkumab subcutaneous (SC) injection at weeks 0, 4, and 12 during placebo-controlled period. At Week 16 participants were crossed over to receive guselkumab 100 milligram (mg) at weeks 16, 20, and 28.
- Guselkumab: Participants received guselkumab 100 mg SC injection at weeks 0, 4, 12, 20 and 28. Participants received placebo at Week 16 to maintain the study blind.
- Placebo to Guselkumab: Participants who received placebo during placebo controlled period was crossed over to receive guselkumab 100 mg SC injection at weeks 16, 20 and 28.
Period: Placebo Controlled Period(Week[wk] 0-16)
Arm/Group | Placebo | Guselkumab | Placebo to Guselkumab
Started | 16 | 62 | 0
Completed | 13 | 61 | 0
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Active Treatment and Follow up (wk16-40)
Arm/Group | Placebo | Guselkumab | Placebo to Guselkumab
Started | 0 | 61 | 13
Completed | 0 | 53 | 13
Not Completed | 0 | 8 | 0
Not completed — Other | 0 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab | Total
Number analyzed (Participants) | 16 | 62 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (15.7) | 46.2 (12.92) | 46 (13.43)
Age, Customized [Count of Participants; unit: Participants]
  >=18 to 65 years | 14 | 58 | 72
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 21 | 25
  Male | 12 | 41 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 60 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 57 | 70
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 3 | 5
  Black or African American | 1 | 1 | 2
  Hispanic or Latino | 0 | 2 | 2
  Other | 0 | 1 | 1
  White Non-Hispanic | 13 | 55 | 68
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 19 | 24
  Poland | 5 | 20 | 25
  United States | 6 | 23 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16
Description: The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). Participants who achieved an IGA score of cleared (0) or minimal (1) were considered IGA cleared or minimal responders. Non-responder imputation (counted as non-responders) was applied for participants who met treatment failure rules, as well as for remaining missing data after treatment failure. Participants who discontinued study drug due to lack of efficacy, an adverse event (AE) of worsening of psoriasis, or who started a protocol-prohibited medication/therapy during study that could improve psoriasis were considered as treatment failures for the study.
Time Frame: Week 16
Population: Full analysis set (FAS) included all randomized participants who received at least 1 injection of study drug. Participants were analyzed according to the assigned treatment to which they were randomized, regardless of the treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants | 0 | 80.6
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p < 0.001, Fisher Exact

2. Primary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI) 90 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percent (%) to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score. Non-responder imputation (counted as non-responders) was applied for participants who met treatment failure rules, as well as for remaining missing data after treatment failure.
Time Frame: Week 16
Population: FAS included all randomized participants who received at least 1 injection of study drug. Participants were analyzed according to the assigned treatment to which they were randomized, regardless of the treatment they actually received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants | 0 | 75.8
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p < 0.001, Fisher Exact

3. Secondary Outcome: Percentage of Participants Who Achieve an IGA Score of Cleared (0) at Week 16
Description: The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). Participants who achieved an IGA score of cleared (0) were considered IGA cleared responders. Non-responder imputation (counted as non-responders) was applied for participants who met treatment failure rules, as well as for remaining missing data after treatment failure.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants | 0 | 56.5

4. Secondary Outcome: Percentage of Participants Who Achieve a PASI 100 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. Participants with 100% improvement in PASI from baseline (PASI score=0) were considered PASI 100 responders. Non-responder imputation (counted as non-responders) was applied for participants who met treatment failure rules, as well as for remaining missing data after treatment failure.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants | 0 | 50.0

5. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of Mild or Better (Less Than or Equal to [<=] 2) at Week 16
Description: The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). Participants who achieved an IGA score of cleared (0), minimal (1), or mild (2) were considered IGA mild or better responders. Non-responder imputation (counted as non-responders) was applied for participants who met treatment failure rules, as well as for remaining missing data after treatment failure.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants | 0 | 93.5

6. Secondary Outcome: Percentage of Participants Who Achieve a PASI 50 Response and a PASI 75 Response at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. Participants with >=50% and >= 75% improvement in PASI from baseline were considered PASI 50 and PASI 75 responders respectively. Non-responder imputation (counted as non-responders) was applied for participants who met treatment failure rules, as well as for remaining missing data after treatment failure.
Time Frame: Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants
  PASI 50 responders | 0 | 93.5
  PASI 75 responders | 0 | 88.7

7. Secondary Outcome: Percent Improvement From Baseline in PASI Score at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. Participants were analyzed according to the assigned treatment to which they were randomized, regardless of the treatment they actually received.
Time Frame: Baseline and Week 16
Population: FAS included all randomized participants who received at least 1 injection of study drug. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Imputation was applied only for participants who met treatment failure and their missing values were counted as zero.
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 61
Percent improvement | 8.72 (18.229) | 91.53 (16.756)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Percent Improvement From Baseline in PASI Score Through Week 40
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. Participants were analyzed according to the assigned treatment to which they were randomized, regardless of the treatment they actually received. From week 20, participants in placebo group, only included participants who crossed over to receive guselkumab at week 16.
Time Frame: Baseline, Week 4, 8, 12, 20, 24, 28, 32, and Week 40 (4 weeks beyond the recommended every 8 weeks [q8w] dosing interval)
Population: FAS included all randomized participants who received at least 1 injection of study drug. Here, n (number analyzed) signifies number of participants who were analyzed at specific timepoint, for each arm, respectively. Imputation was applied only for participants who met treatment failure and their missing values were counted as zero.
Measure: Mean (Standard Deviation); unit: Percent improvement
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percent improvement
  Week 4 | 5.58 (13.970) | 40.99 (26.377)
  Week 8 | 10.45 (21.540) | 71.76 (26.984)
  Week 12: number analyzed (Participants) | 16 | 61
  Week 12 | 13.76 (24.143) | 84.97 (20.520)
  Week 20: number analyzed (Participants) | 13 | 61
  Week 20 | 62.65 (20.760) | 94.77 (13.179)
  Week 24: number analyzed (Participants) | 13 | 59
  Week 24 | 88.74 (12.092) | 95.89 (10.164)
  Week 28: number analyzed (Participants) | 13 | 60
  Week 28 | 95.68 (6.162) | 96.30 (7.504)
  Week 32: number analyzed (Participants) | 13 | 58
  Week 32 | 96.16 (5.602) | 96.64 (7.143)
  Week 40: number analyzed (Participants) | 13 | 55
  Week 40 | 97.70 (3.443) | 92.47 (13.289)

9. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of Cleared (0), Cleared (0) or Minimal (1) and Mild or Better (<=2) Through Week 40
Description: The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). Participants who achieved an IGA score of cleared (0) or minimal (1) were considered IGA cleared or minimal responders while those achieved an IGA score of cleared (0), minimal (1), or mild (2) were considered IGA mild or better responders. Participants were analyzed according to the assigned treatment to which they were randomized, regardless of the treatment they actually received. From week 20, participants in placebo group, only included participants who crossed over to receive guselkumab at week 16.
Time Frame: Week 4, 8, 12, 20, 24, 28, 32, and Week 40 (4 weeks beyond the recommended q8w dosing interval)
Population: FAS included all randomized participants who received at least 1 injection of study drug. Here, n (number analyzed) signifies number of participants who were analyzed at specific timepoint, for each arm, respectively. Non-responder imputation was used to impute missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants
  Week 4: IGA of cleared (0) | 0 | 4.8
  Week 4: IGA of cleared (0) or minimal (1) | 0 | 19.4
  Week 4: IGA of mild or better (<=2) | 0 | 54.8
  Week 8: IGA of cleared (0) | 0 | 19.4
  Week 8: IGA of cleared (0) or minimal (1) | 0 | 56.5
  Week 8: IGA of mild or better (<=2) | 12.5 | 85.5
  Week 12: IGA of cleared (0) | 0 | 35.5
  Week 12: IGA of cleared (0) or minimal (1) | 0 | 67.7
  Week 12: IGA of mild or better (<=2) | 0 | 91.9
  Week 20: IGA of cleared (0): number analyzed (Participants) | 13 | 62
  Week 20: IGA of cleared (0) | 0 | 67.7
  Week 20: IGA of cleared (0) or minimal (1): number analyzed (Participants) | 13 | 62
  Week 20: IGA of cleared (0) or minimal (1) | 46.2 | 85.5
  Week 20: IGA of mild or better (<=2): number analyzed (Participants) | 13 | 62
  Week 20: IGA of mild or better (<=2) | 92.3 | 93.5
  Week 24: IGA of cleared (0): number analyzed (Participants) | 13 | 62
  Week 24: IGA of cleared (0) | 38.5 | 71.0
  Week 24: IGA of cleared (0) or minimal (1): number analyzed (Participants) | 13 | 62
  Week 24: IGA of cleared (0) or minimal (1) | 100.0 | 87.1
  Week 24: IGA of mild or better (<=2): number analyzed (Participants) | 13 | 62
  Week 24: IGA of mild or better (<=2) | 100.0 | 88.7
  Week 28: IGA of cleared (0): number analyzed (Participants) | 13 | 62
  Week 28: IGA of cleared (0) | 61.5 | 64.5
  Week 28: IGA of cleared (0) or minimal (1): number analyzed (Participants) | 13 | 62
  Week 28: IGA of cleared (0) or minimal (1) | 100.0 | 87.1
  Week 28: IGA of mild or better (<=2): number analyzed (Participants) | 13 | 62
  Week 28: IGA of mild or better (<=2) | 100.0 | 95.2
  Week 32: IGA of cleared (0): number analyzed (Participants) | 13 | 62
  Week 32: IGA of cleared (0) | 69.2 | 66.1
  Week 32: IGA of cleared (0) or minimal (1): number analyzed (Participants) | 13 | 62
  Week 32: IGA of cleared (0) or minimal (1) | 92.3 | 82.3
  Week 32: IGA of mild or better (<=2): number analyzed (Participants) | 13 | 62
  Week 32: IGA of mild or better (<=2) | 100.0 | 90.3
  Week 40: IGA of cleared (0): number analyzed (Participants) | 13 | 62
  Week 40: IGA of cleared (0) | 61.5 | 53.2
  Week 40: IGA of cleared (0) or minimal (1): number analyzed (Participants) | 13 | 62
  Week 40: IGA of cleared (0) or minimal (1) | 92.3 | 71.0
  Week 40:IGA of mild or better (<=2): number analyzed (Participants) | 13 | 62
  Week 40:IGA of mild or better (<=2) | 100.0 | 79.0

10. Secondary Outcome: Percentage of Participants Who Achieved PASI 100 Responses, PASI 90 Responses, PASI 75 Responses, and PASI 50 Responses
Description: PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In PASI system, body is divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. PASI produces a numeric score that can range from 0 (no psoriasis) to 72.Participants with >=50%, >= 75%, >=90% and >= 100% improvement in PASI from baseline were considered PASI 50, 75, 90 and PASI 100 responders, respectively. Participants were analyzed according to the assigned treatment to which they were randomized, regardless of the treatment they actually received. From week 20, participants in placebo group, only included participants who crossed over to receive guselkumab at week 16.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 32, and Week 40 (4 weeks beyond the recommended q8w dosing interval)
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 62
Percentage of participants
  Week 4: 100% improvement | 0 | 3.2
  Week 4: >= 90% improvement | 0 | 4.8
  Week 4: >= 75% improvement | 0 | 12.9
  Week 4: >= 50% improvement | 0 | 33.9
  Week 8: 100% improvement | 0 | 16.1
  Week 8: >= 90% improvement | 0 | 33.9
  Week 8: >= 75% improvement | 0 | 56.5
  Week 8: >= 50% improvement | 6.3 | 80.6
  Week 12: 100% improvement | 0 | 30.6
  Week 12: >= 90% improvement | 0 | 54.8
  Week 12: >= 75% improvement | 0 | 77.4
  Week 12: >= 50% improvement | 12.5 | 90.3
  Week 16: 100% improvement | 0 | 50.0
  Week 16: >=90% improvement | 0 | 75.8
  Week 16: >=75% improvement | 0 | 88.7
  Week 16: >=50% improvement | 0 | 93.5
  Week 20: 100% improvement: number analyzed (Participants) | 13 | 62
  Week 20: 100% improvement | 0 | 66.1
  Week 20: >=90% improvement: number analyzed (Participants) | 13 | 62
  Week 20: >=90% improvement | 7.7 | 85.5
  Week 20: >=75% improvement: number analyzed (Participants) | 13 | 62
  Week 20: >=75% improvement | 30.8 | 91.9
  Week 20: >=50% improvement: number analyzed (Participants) | 13 | 62
  Week 20: >=50% improvement | 69.2 | 95.2
  Week 24: 100% improvement: number analyzed (Participants) | 13 | 62
  Week 24: 100% improvement | 30.8 | 71.0
  Week 24: >=90% improvement: number analyzed (Participants) | 13 | 62
  Week 24: >=90% improvement | 61.5 | 82.3
  Week 24: >=75% improvement: number analyzed (Participants) | 13 | 62
  Week 24: >=75% improvement | 84.6 | 88.7
  Week 24: >=50% improvement: number analyzed (Participants) | 13 | 62
  Week 24: >=50% improvement | 100.0 | 95.2
  Week 28: 100% improvement: number analyzed (Participants) | 13 | 62
  Week 28: 100% improvement | 53.8 | 64.5
  Week 28: >=90% improvement: number analyzed (Participants) | 13 | 62
  Week 28: >=90% improvement | 84.6 | 85.5
  Week 28: >=75% improvement: number analyzed (Participants) | 13 | 62
  Week 28: >=75% improvement | 100.0 | 95.2
  Week 28: >50% improvement: number analyzed (Participants) | 13 | 62
  Week 28: >50% improvement | 100.0 | 96.8
  Week 32: 100% improvement: number analyzed (Participants) | 13 | 62
  Week 32: 100% improvement | 61.5 | 64.5
  Week 32: >=90% improvement: number analyzed (Participants) | 13 | 62
  Week 32: >=90% improvement | 84.6 | 85.5
  Week 32: >=75% improvement: number analyzed (Participants) | 13 | 62
  Week 32: >=75% improvement | 100.0 | 90.3
  Week 32: >=50% improvement: number analyzed (Participants) | 13 | 62
  Week 32: >=50% improvement | 100.0 | 93.5
  Week 40: 100% improvement: number analyzed (Participants) | 13 | 62
  Week 40: 100% improvement | 53.8 | 53.2
  Week 40: >=90% improvement: number analyzed (Participants) | 13 | 62
  Week 40: >=90% improvement | 100.0 | 66.1
  Week 40: >=75% improvement: number analyzed (Participants) | 13 | 62
  Week 40: >=75% improvement | 100.0 | 79.0
  Week 40: >=50% improvement: number analyzed (Participants) | 13 | 62
  Week 40: >=50% improvement | 100.0 | 79.0

ADVERSE EVENTS:
Time Frame: Up to Week 40
Groups:
- Placebo (Week 0-16): Participants received placebo matched to guselkumab subcutaneous (SC) injection at weeks 0, 4, and 12 during placebo-controlled period. At Week 16 participants were crossed over to receive guselkumab 100 milligram (mg) at weeks 16, 20, and 28.
- Guselkumab (Week 0-16): Participants received guselkumab 100 mg SC injection at weeks 0, 4, 12, 20 and 28. Participants received placebo at Week 16 to maintain the study blind.
- Placebo to Guselkumab (Week 16-40): Participants who received placebo during placebo controlled period was crossed over to receive guselkumab 100 mg SC injection at weeks 16, 20 and 28.
- Guselkumab (Week 16-40): Participants received placebo at Week 16, and 100 mg guselkumab at Week 20 and 28.
Arm/Group | Placebo (Week 0-16) | Guselkumab (Week 0-16) | Placebo to Guselkumab (Week 16-40) | Guselkumab (Week 16-40)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/62 | 0/13 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/62 | 2/13 | 1/61
Other Adverse Events (participants affected / at risk) | 12/16 | 38/62 | 8/13 | 24/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-16) (N=16) | Guselkumab (Week 0-16) (N=62) | Placebo to Guselkumab (Week 16-40) (N=13) | Guselkumab (Week 16-40) (N=61)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-16) (N=16) | Guselkumab (Week 0-16) (N=62) | Placebo to Guselkumab (Week 16-40) (N=13) | Guselkumab (Week 16-40) (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Injection Site Bruising (General disorders) | 1 | 2 | 1 | 1
Injection Site Coldness (General disorders) | 3 | 14 | 2 | 7
Injection Site Erythema (General disorders) | 1 | 7 | 0 | 4
Injection Site Induration (General disorders) | 2 | 7 | 1 | 2
Injection Site Oedema (General disorders) | 1 | 0 | 0 | 0
Injection Site Pain (General disorders) | 7 | 25 | 3 | 11
Injection Site Pruritus (General disorders) | 2 | 8 | 1 | 2
Injection Site Swelling (General disorders) | 1 | 7 | 1 | 3
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 5 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3 | 1 | 6
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Urticaria Pressure (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT02905331/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT02905331/SAP_001.pdf